CLINICAL TRIAL: NCT05728476
Title: Microinvasive Pars Plana Vitrectomy Combined ILM Peeling Versus Anti-VEGF Intravitreal Injection for Treatment-naïve Diabetic Macular Edema
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Eye Hospital (Other)
Responsible Party: Principal Investigator, Bojie Hu, Professor, Tianjin Medical University Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TianjinMUEHhbj111
Record Dates: First submitted 2023-02-02; First posted 2023-02-15 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2023-10

CONDITIONS: Diabetic Macular Edema; Pars Plana Vitrectomy; Conbercept
MeSH Terms: interventions — KH902 fusion protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitrectomy group (Experimental): Standard 25-gauge PPV will be performed by an experienced surgeon under retrobulbar anesthesia. After clearing the central vitreous, a complete posterior vitreous detachment (PVD) will be achieved with aspiration to remove the tightly attached posterior hyaloid. The vitreous will be removed by a high-speed vitrectomy surgical system (Constellation Vision System, Alcon Laboratories, Fort Worth, Texas, USA). The ILM stained with indocyanine green (ICG) will be peeled up to the vascular arcades. In case of need, panretinal photocoagulation (PRP) can be performed during surgery. The vitreous cavity will be filled with balanced salt solution (BSS) at the end of the procedure.
  Interventions: Procedure: Vitrectomy combined with ILM peeling
- Anti-VEGF group (Active Comparator): Patients will receive three monthly intravitreal injections of 0.5 mg Conbercept (Chengdu Kanghong Biotech Co.) with a 30-gauge syringe needle approximately 3.5-4 mm posterior to the corneal limbus under topical anesthesia.
  Interventions: Drug: Conbercept intravitreal injection

INTERVENTIONS:
Procedure: Vitrectomy combined with ILM peeling — Standard 25-gauge PPV will be performed by an experienced surgeon under retrobulbar anesthesia. After clearing the central vitreous, a complete posterior vitreous detachment (PVD) will be achieved with aspiration to remove the tightly attached posterior hyaloid. The vitreous will be removed by a high-speed vitrectomy surgical system (Constellation Vision System, Alcon Laboratories, Fort Worth, Texas, USA). The ILM stained with indocyanine green (ICG) will be peeled up to the vascular arcades. In case of need, panretinal photocoagulation (PRP) can be performed during surgery. The vitreous cavity will be filled with balanced salt solution (BSS) at the end of the procedure.
  Arms: Vitrectomy group
Drug: Conbercept intravitreal injection — Patients will receive three monthly intravitreal injections of 0.5 mg Conbercept (Chengdu Kanghong Biotech Co.) with a 30-gauge syringe needle approximately 3.5-4 mm posterior to the corneal limbus under topical anesthesia.
  Arms: Anti-VEGF group

SUMMARY:
Diabetic macular edema (DME) is the main cause of vision loss in patients with diabetes. At present, anti-vascular endothelial growth factor (VEGF) intravitreal injection is the first-line therapy for DME, nevertheless, some patients do not respond well to anti-VEGF agents and often require multiple injections, which increases the psychological and economic burden of patients. Microinvasive pars plana vitrectomy (PPV) has been proven to be safe and effective for refractory DME. However, there are few studies on treatment-naïve DME. The purpose of this study is to explore whether early PPV combined with internal limiting membrane (ILM) peeling can reduce the treatment burden of DME patients, prevent vision loss, and maintain long-term stabilization of diabetic retinopathy.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Patients and their families fully understand the research and sign the informed consent form
* Diagnosed with type 1 or 2 diabetes mellitus
* Hemoglobin A1c (HbA1c) of less than 10% within 3 months
* Clear media for adequate OCT and optical coherence tomography angiography (OCTA) images
* Treatment-naïve DME diagnosed clinically
* Central subfield thickness (CST) of >300μm and intra- or subretinal fluid seen on (spectral-domain) SD-OCT
* Early Treatment Diabetic Retinopathy Study (ETDRS) BCVA between 24 and 73 letters on the day of randomization
* Treatment within 12 months of DME diagnosis
* No contraindication of vitrectomy or conbercept intravitreal injection

Exclusion Criteria:

* Any previous DME treatment (i.e. anti-VEGF injections, intraocular corticosteroids, macular photocoagulation)
* Macular edema caused by other disease (i.e. neovascular age-related macular degeneration, retinal vein occlusion, uveitis)
* Any previous intraocular surgeries (cataract surgery performed at least 3 months before study entry will not be exclusionary)
* Vision loss caused by other ocular disease (i.e. cataract, proliferative diabetic retinopathy, glaucoma, high myopia)
* A follow-up duration of less than 12 months
* Severe dysfunction of the heart, liver, kidney, lung and other organs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-09-05 (Estimated); Study Completion 2026-09-05 (Estimated)

PRIMARY OUTCOMES:
Best corrected visual acuity change (BCVA) | 1, 3, 6, 12 month postoperatively
  Early Treatment Diabetic Retinopathy Study (ETDRS) Alphabet Chart
Central subfield thickness (CST) change | 1, 3, 6, 12 month postoperatively
  Three-dimensional spectral domain optical coherence tomography (SD-OCT)

SECONDARY OUTCOMES:
The stage of diabetic retinopathy (DR) | 12 month postoperatively
  The grading and classification of DR will follow the International Clinical Diabetic Retinopathy and Diabetic Macular Oedema Disease Severity Scales. Ultra-wide field fundus photography will help investigators grade diabetic retinopathy.
Cost-effectiveness analysis | 12 month postoperatively
  The incremental cost-effectiveness ratio (ICER) is used as the evaluation index in cost-effectiveness analysis. The average cost of the two groups of treatments is taken as willingness to pay (WTP). If ICER is less than WTP, the treatment scheme is cost-effective.
Vision-related quality of life questionnaire | 6, 12 month postoperatively
  The National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) will be used to evaluate the vision-related quality of life. Scores range from 0 to 100, and lower scores indicate a poorer quality of life.
Biomarkers of optical coherence tomography (OCT) | 1, 3, 6, 12 month postoperatively
  Scanning was centred on the macular fovea with a scan length of 6 mm. The resolution was 5 μm, the scan depth was 4 mm, and the scan mode was horizontal linear scanning of 512×128.
Biomarkers of OCT angiography (OCTA) | 1, 3, 6, 12 month postoperatively
  The scanning area, centred on the fovea, was captured in 3×3 mm sections with a resolution of 304×304 pixels.
Occurrence rates of re-treatment | 12 months postoperatively
  Pro re nata conbercept treatment will be performed if the following criteria are met: (1) existence of recent or persisting cystoid retinal lesions; (2) a decrease of no less than 5 ETDRS letters in BCVA; and (3) an increase of 50 μm or more in CST compared with the best value previously achieved.
Occurrence rates of adverse events | 12 months postoperatively
  Ocular hypertension, progression of cataract, corneal abrasion, retinal injury, hyphaemia, uveitis or inflammatory reaction, and endophthalmitis.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Guo H, Li W, Nie Z, Zhang X, Jiao M, Bai S, Duan N, Li X, Hu B. Microinvasive pars plana vitrectomy combined with internal limiting membrane peeling versus anti-VEGF intravitreal injection for treatment-naive diabetic macular edema (VVV-DME study): study protocol for a randomized controlled trial. Trials. 2023 Oct 24;24(1):685. doi: 10.1186/s13063-023-07735-w. PMID 37875997